CLINICAL TRIAL: NCT07106086
Title: Combined Effect of Scapulothoracic Mobilization With Buteyko Breathing on Pulmonary Parameters Functional Capacity and Balance Among COPD (Chronic Obstructive Pulmonary Disease) Patients
Brief Title: Combined Effect of Scapulothoracic Mobilization With Buteyko Breathing on COPD (Chronic Obstructive Pulmonary Disease) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rashid Latif Medical College (Other)
Responsible Party: Principal Investigator, Aleena Waheed, Physiotherapist, Rashid Latif Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB/2023/130
Record Dates: First submitted 2025-07-28; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Balance; Breathing; COPD; Functional Capacity; Mobilization
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scapulothoracic mobilization with buteyko breathing (Experimental): Scapulothoracic mobilization with buteyko breathing
  Interventions: Other: Scapulothoracic mobilization; Other: Buteyko breathing
- Buteyko breathing (Active Comparator): buteyko breathing
  Interventions: Other: Buteyko breathing

INTERVENTIONS:
Other: Scapulothoracic mobilization — Scapulothoracic Mobilization and Buteyko Breathing Technique:
  Subjects lay supine with arms crossed, hands on opposite scapulae. The interventionist stabilized elbows and applied pressure to shoulders, with one hand on the spine using a loose fist to mobilize vertebrae. Various spinal motions-rotation, flexion, lateral flexion, and translation-were assessed. In a lateral position, the subject bent both knees and placed the upper arm on a cushion. The interventionist stood close, placing fingers under the scapula's medial border.
  Arms: Scapulothoracic mobilization with buteyko breathing
Other: Buteyko breathing — Buteyko Breathing: Subjects sat upright, relaxed respiratory muscles, and breathed gently through the nose. The sequence included calm nasal inhalation and exhalation using the diaphragm, followed by shallow inhalation and slow exhalation. A brief post-exhalation breath hold was added. The cycle was repeated for several minutes.

SUMMARY:
The objective of this study will be to determine the combine effect of scapulothoracic mobilization with Buteyko breathing on pulmonary parameters functional capacity and balance among COPD patient.

DETAILED DESCRIPTION:
The study will be Randomized Clinical Trial which include forty (40) subjects clinically diagnosed according to Global Initiative for Obstructive Lung Disease (GOLD) standard of chronic obstructive pulmonary disease (COPD). Patients will be allocated into two groups i.e. Group A (20) and Group B (20). Group A scapulothoracic mobilization with Buteyko breathing (BBT) and Group B received Buteyko breathing (BBT). The Pulse oximeter will be used to evaluate Pulmonary parameters. The 6-meter walk test will be used to assess functional capacity. The Activities-specific balance confidence scale (ABC scale) will be used to assess Balance Confidence and Single leg stance (SLS) will be used to evaluate balance. The evaluation will be done on day one as pretreatment values and post-treatment values at the end of third week.

ELIGIBILITY:
Inclusion Criteria:

* Clinically Diagnosed COPD is confirmed by diagnostic criteria of COPD (forced expiratory volume in 1 second [FEV1] <80% predicted, FEV1/forced vital capacity [FVC] <0.7 predicted) according to the international guideline and the ability to provide inform consent.
* Patients with Resting Respiratory Rate >_ 24

Exclusion Criteria

* Patients diagnosed with a primary pulmonary vascular disease
* Patients diagnosed with severe psychiatric disorders and cognitive dysfunction
* Patients diagnosed severe auditory/visual impairments
* Patients diagnosed Musculoskeletal, Rheumatic ,Cardiac/Neurological disorder and Malignancies
* Patients diagnosed with skin, peripheral vascular disorder excluded

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-07-20 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Oxygen Saturation | Pre and 2 week Post intervention
  Oxygen saturation is measured by Pulse oximeter The gold standard for measuring arterial blood oxygen saturation (SaO₂) requires arterial blood sampling, but pulse oximetry provides a non-invasive estimate (SpO₂) widely used to detect hypoxemia.
Functional capacity | Pre and 2 week post intervention
  Functional Capacity is measured by 6- minute walk test. The 6-minute walk test (6MWT) is a well-known tool to measure ability to walk and endurance in the sub-maximal condition. The 6MWT is a exercise test that involves measuring the distance walked over a span of 6 minutes. Participants were encouraged to walk on a straight, flat surface as fast as possible for 6 minutes on a marked course, with pauses as necessary.
Balance | Pre and 2 week post intervention
  The Balance is measured by Single leg stance test. Single Leg Stance (SLS). The SLS is a simple balance test where the participant stands on one leg for as long as possible (up to 60 seconds) with hands on hips. The test is performed first with eyes open, then with eyes closed. Longer duration indicates better balance. The SLS has demonstrated excellent reliability in individuals with COPD as well as in community-dwelling older adults.

SECONDARY OUTCOMES:
Respiratory rate | Pre and Post 2 week intervention
  Respiratory rate is measured by Pulse oximeter Pulse oximetry can reliably estimate respiratory rate (RR) and is suitable for wearable use due to its compactness and cost-effectiveness.
Heart rate | Pre and Post 2 week intervention
  Heart rate is measured by the Pulse oximeter. Normal resting heart rate ranges from 60-100 bpm, but it may fluctuate. COPD patients often show elevated resting HR. Pulse oximeters can effectively monitor HR.

CONTACTS AND LOCATIONS:
Locations (1):
- Arif Memorial Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Not Decided yet

REFERENCES:
- [Background] Jarhyan P, Hutchinson A, Khaw D, Prabhakaran D, Mohan S. Prevalence of chronic obstructive pulmonary disease and chronic bronchitis in eight countries: a systematic review and meta-analysis. Bull World Health Organ. 2022 Mar 1;100(3):216-230. doi: 10.2471/BLT.21.286870. Epub 2022 Jan 19. PMID 35261410
- [Background] Gore S, Blackwood J, Ziccardi T. Associations Between Cognitive Function, Balance, and Gait Speed in Community-Dwelling Older Adults with COPD. J Geriatr Phys Ther. 2023 Jan-Mar 01;46(1):46-52. doi: 10.1519/JPT.0000000000000323. Epub 2021 Jul 29. PMID 34334706
- [Background] Chen Y, Li P, Wang J, Wu W, Liu X. Assessments and Targeted Rehabilitation Therapies for Diaphragmatic Dysfunction in Patients with Chronic Obstructive Pulmonary Disease: A Narrative Review. Int J Chron Obstruct Pulmon Dis. 2022 Mar 3;17:457-473. doi: 10.2147/COPD.S338583. eCollection 2022. PMID 35273448
- [Background] Berriet AC, Beaumont M, Peran L, Le Ber C, Couturaud F. Effects of pulmonary rehabilitation on fear of falling in Chronic Obstructive Pulmonary Disease (COPD) patients: An observational study. Respir Med Res. 2022 Nov;82:100932. doi: 10.1016/j.resmer.2022.100932. Epub 2022 Jun 12. PMID 35878569
- [Background] Alqahtani JS. Prevalence, incidence, morbidity and mortality rates of COPD in Saudi Arabia: Trends in burden of COPD from 1990 to 2019. PLoS One. 2022 May 19;17(5):e0268772. doi: 10.1371/journal.pone.0268772. eCollection 2022. PMID 35588429
- [Background] Agusti A, Celli BR, Criner GJ, Halpin D, Anzueto A, Barnes P, Bourbeau J, Han MK, Martinez FJ, Montes de Oca M, Mortimer K, Papi A, Pavord I, Roche N, Salvi S, Sin DD, Singh D, Stockley R, Lopez Varela MV, Wedzicha JA, Vogelmeier CF. Global Initiative for Chronic Obstructive Lung Disease 2023 Report: GOLD Executive Summary. Eur Respir J. 2023 Apr 1;61(4):2300239. doi: 10.1183/13993003.00239-2023. Print 2023 Apr. PMID 36858443